CLINICAL TRIAL: NCT04341116
Title: A Phase 2/3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of TJ003234 in Subjects With Severe Coronavirus Disease 2019 (COVID-19)
Brief Title: Study of TJ003234 (Anti-GM-CSF Monoclonal Antibody) in Subjects With Severe Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: I-Mab Biopharma US Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJ003234COV201
Record Dates: First submitted 2020-04-04; First posted 2020-04-10 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Coronavirus Disease 2019 COVID-19
MeSH Terms: interventions — plonmarlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TJ003234 Medium Dose (Experimental)
  Interventions: Drug: TJ003234
- TJ003234 Low Dose (Experimental): Part 1 only
  Interventions: Drug: TJ003234
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TJ003234 High Dose (Experimental): Part 2 Phase 3 only
  Interventions: Drug: TJ003234

INTERVENTIONS:
Drug: TJ003234 — patients receive a single infusion
  Arms: TJ003234 High Dose; TJ003234 Low Dose; TJ003234 Medium Dose
Drug: Placebo — patients receive a single infusion
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center trial to evaluate the safety and efficacy of TJ003234 administered as an intravenous (IV) infusion in subjects with severe COVID-19 under supportive care, and to assess the effect of TJ003234 on the levels of cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older (including 18 years); male or female
* Laboratory-confirmed SARS-CoV-2 or COVID-19 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay.
* Bilateral lung infection confirmed by imaging.
* Severe disease that meets one of the following conditions: (i) At rest, finger blood oxygen saturation ≤ 93% or PaO2/FiO2 ≤ 300 mmHg; (ii) Requiring non-invasive or invasive mechanical ventilation; OR (iii) Requiring high flow oxygen ≥ 15L/min
* Hospitalized for no more than 5 calendar days at the time of screening

Exclusion Criteria:

* Any previous and/or current clinically significant disease or condition that has not been stable within 3 months prior to enrollment, or acute illness, planned medical/ surgical procedure, or any trauma that occurred within 2 weeks prior to enrollment.
* Chronic obstructive pulmonary disease (COPD) patients requiring inhaled corticosteroid, long-acting beta-adrenergic agonists, long-acting anticholinergics, or long-term oxygen therapy (Part 1 only).
* Pulmonary interstitial disease, pulmonary alveolar proteinosis, and pulmonary granulomatosis.
* Cardiovascular event in the 3 months prior to study drug administration: acute myocardial infarction or unstable angina pectoris, severe arrhythmia (multiple sources of frequent ventricular premature beat, ventricular tachycardia and ventricular fibrillation); New York Heart Association Classification (NYHA): Class III-Class IV.
* Blood system disorders or routine blood analysis test abnormalities: Hemoglobin < 8 g/dL; Absolute neutrophil count (ANC) <1500 × 109/L; Platelets < 50 × 109/L.
* Dependence on glucocorticoid treatment equivalent to methylprednisolone 2 mg/kg/ day or more or long-term use of anti-rejection or immunomodulatory drugs.
* Subjects that have been on invasive mechanical ventilation for ≥120 hours at the time of dosing
* Subjects that require ECMO.
* Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Xu, MD, PhD, Study Director — I-Mab Biopharma US Limited
Locations (14):
- United States (14):
  - University of Arkansas, Little Rock, Arkansas
  - Olive View-UCLA Medical Center, Sylmar, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - OSF Healthcare Saint Francis Medical Center, Peoria, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Medpharmics, LLC, Metairie, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - UNM Hospitals, Albuquerque, New Mexico
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- TJ003234 3mg/kg (Part 1): Subjects treated with 3mg/kg of TJ003234
- TJ003234 6mg/kg (Part 1): Subjects treated with 6mg/kg TJ003234
- Placebo (Part 1): Subjects treated with placebo in Part 1
- TJ003234 6mg/kg (Part 2): Subjects treated with 6mg/kg in Part 2
- TJ003234 10mg/kg (Part 2): Subjects treated with 10mg/kg of TJ003234
- Placebo (Part 2): Subjects treated with placebo in Part 2
Period: Overall Study
Arm/Group | TJ003234 3mg/kg (Part 1) | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6mg/kg (Part 2) | TJ003234 10mg/kg (Part 2) | Placebo (Part 2)
Started | 8 | 8 | 8 | 77 (ITT population) | 6 | 42 (ITT population)
Completed | 7 | 6 | 6 | 66 | 5 | 34
Not Completed | 1 | 2 | 2 | 11 | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- TJ003234 3mg/kg (Part 1): subjects treated by 3mg/kg of TJ003234
- TJ003234 6mg/kg (Part 1): subjects treated by 6mg/kg of TJ003234 in Part 1
- Placebo (Part 1): subjects treated by placebo in Part 1
- TJ003234 6mg/kg (Part 2): subjects treated by 6mg/kg of TJ003234 in Part 2
- TJ003234 10mg/kg (Part 2): subjects treated by 10 mg/kg of TJ003234 in Part 2
- Placebo (Part 2): subjects treated by placebo in Part 2
- Total: Total of all reporting groups
Arm/Group | TJ003234 3mg/kg (Part 1) | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6mg/kg (Part 2) | TJ003234 10mg/kg (Part 2) | Placebo (Part 2) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 77 | 6 | 42 | 149
Age, Continuous [Mean (Full Range); unit: years] | 51.9 [36 to 80] | 58.4 [39 to 75] | 58 [19 to 80] | 55.6 [24 to 84] | 57.2 [31 to 75] | 56.4 [37 to 77] | 56 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 49 | 4 | 24 | 88
  Male | 4 | 5 | 4 | 28 | 2 | 18 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 33 | 2 | 16 | 53
  Not Hispanic or Latino | 8 | 7 | 7 | 44 | 4 | 26 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 4 | 3 | 3 | 23 | 3 | 10 | 46
  White | 4 | 5 | 5 | 39 | 3 | 21 | 77
  More than one race | 0 | 0 | 0 | 11 | 0 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 77 | 6 | 42 | 149
Height [Mean (Full Range); unit: cm] | 168.8 [144.8 to 190.5] | 166.8 [147.3 to 185.4] | 173.3 [160.0 to 190.5] | 167.1 [72.0 to 190.5] | 171.0 [160.0 to 182.9] | 168.3 [149.9 to 188.0] | 168.65 [72.0 to 190.5]
Weight [Mean (Full Range); unit: kg] | 101.4 [43.9 to 161.0] | 88.0 [74.0 to 138.3] | 108.9 [53.0 to 145.0] | 97.2 [43.9 to 161.0] | 98.1 [74.0 to 138.3] | 97.1 [53.0 to 145.0] | 98.3 [43.9 to 161.0]
Mechanical Ventilation [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 3 | 10 | 0 | 6 | 25
  No | 3 | 1 | 2 | 67 | 6 | 36 | 115
  Unknown | 2 | 4 | 3 | 0 | 0 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Alive and Free of Mechanical Ventilation Among Subjects Who Are Free of Mechanical Ventilation at Baseline
Description: Free of mechanical ventilation was defined as proportion of subjects who scores 1 to 5 in the following 8-category ordinal scale.
  8, death; 7, ventilation in addition to extracorporeal membrane oxygen (ECMO), continuous renal replacement therapy (CRRT) or pressors; 6, intubation and mechanical ventilation; 5, non-invasive mechanical ventilation (NIV) or high-flow oxygen; 4, hospitalization with oxygen by mask or nasal prongs; 3. Hospitalization without oxygen supplementation; 2, limitation of activities, discharge from hospital; and 1, no limitation of activities, discharge from hospital.
Time Frame: Day 1 through Day 30
Population: All subjects randomized to treatment who were mechanical ventilation free at baseline was collected only for Part 2 arms/groups. Data was not collected from the Part 1 Arms/Groups.
Measure: Count of Participants; unit: Participants
Groups:
- TJ003234 6mg/kg (Part 1): subjects treated with TJ003234 6mg/kg -Part 1
- Placebo (Part 1): subjects treated with placebo (Part 1)
- TJ003234 6mg/kg (Part 2): subjects treated with TJ003234 6mg/kg (mITT population)
- TJ0032034 10mg/kg (Part 2): subjects treated with TJ003234 10mg/kg (mITT population)
- Placebo (Part 2): Subjects treated with placebo (mITT population)
Arm/Group | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6mg/kg (Part 2) | TJ0032034 10mg/kg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 0 | 0 | 67 | 6 | 36
Participants |  |  | 56 | 5 | 27
Statistical Analysis 1: Comparison: TJ003234 6mg/kg (Part 2) vs TJ0032034 10mg/kg (Part 2); Test type: Superiority; p = .28, Fisher Exact; Median Difference (Final Values) = 9, 95% CI 2-sided [-6.5 to 27], Standard Error of Mean 8.5

2. Secondary Outcome: Percentage of Recovery by Day 14
Description: Sustained recovery in clinical status was defined as patients who have hospitalization without oxygen supplement or discharge from hospital.
Time Frame: Day 1 through Day 14
Population: All subjects randomized was collected only for Part 2 arms/groups. Data was not collected from the Part 1 Arms/Groups.
Measure: Count of Participants; unit: Participants
Groups:
- TJ003234 6mg/kg (Part 1): subjects treated with TJ003234 6mg/kg part 1
- TJ003234 6mg/kg (Part 2): subjects treated with 6mg/kg TJ003234-(ITT population)
- TJ003234 10mg/kg (Part 2): subjects treated10mg/kg TJ003234 (ITT population)
- Placebo (Part 2): Subjects who were treated with Placebo (ITT population)
Arm/Group | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6mg/kg (Part 2) | TJ003234 10mg/kg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 0 | 0 | 77 | 6 | 42
Participants |  |  | 47 | 5 | 20

3. Secondary Outcome: Percentage of Subjects Recovered on Day 30
Description: as for outcome 2
Time Frame: Day 1 through Day 30
Population: All subjects randomized was collected only for Part 2 arms/groups. Data was not collected from the Part 1 Arms/Groups.
Measure: Count of Participants; unit: Participants
Groups:
- TJ003234 6mg/kg (Part 1): subjects treated with 6mg/kg part 1
- Placebo (Part 1): subjects treated with placebo part 1
- TJ003234 6mg/kg (Part 2): subjects treated with 6mg/kg TJ003234 (ITT population)
- TJ003234 10mg/kg (Part 2): subjects treated with 10mg/kg placebo- ITT population
- Placebo (Part 2): subjects treated with placebo-ITT population
Arm/Group | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6mg/kg (Part 2) | TJ003234 10mg/kg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 0 | 0 | 77 | 6 | 42
Participants |  |  | 56 | 5 | 27

4. Secondary Outcome: All-cause Mortality Rate by Day 30
Description: The percentage of subjects who deceased by any cause.
Time Frame: Day 1 through Day 30
Population: All subjects randomized was collected only for Part 2 arms/groups. Data was not collected from the Part 1 Arms/Groups.
Measure: Count of Participants; unit: Participants
Groups:
- TJ003234 6mg/kg (Part 1): subjects treated with TJ003234 6mg/kg - part 1
- Placebo (Part 1): subjects treated with placebo
- TJ003234 6mg/kg (Part 2): subjects treated with 6 mg/kg TJ003234 (ITT population)
- TJ003204 10mg/kg (Part 2): subjects who were treated with 10mg/kg TJ003234 (ITT population)
- Placebo (Part 2): subjects treated by placebo (ITT population)
Arm/Group | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6mg/kg (Part 2) | TJ003204 10mg/kg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 0 | 0 | 77 | 6 | 42
Participants |  |  | 7 | 1 | 9

5. Secondary Outcome: Time to Recovery Among Subjects Alive by Day 30
Description: Time to sustained recovery
Time Frame: Day 1 through Day 30
Population: All subjects randomized without mechanical ventilation Part 2. Part 1 is designed as a randomized, double-blind, placebo-controlled, 3-arm, parallel-group study to evaluate the safety of plonmarlimab in subjects with severe COVID-19. So, no available efficacy data for this part.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- TJ003234 6mg/kg (Part 1): subjects treated with TJ003234 6mg/kg- part 1
- TJ003234 6mg/kg (Part 2): subjects treated with 6mg/kg TJ003234 (mITT population)
- TJ004309 10mg/kg (Part 2): subjects treated with 10mg/kg TJ0032034 (mITT population)
- Placebo (Part 2): subjects treated by placebo (mITT population)
Arm/Group | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6mg/kg (Part 2) | TJ004309 10mg/kg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 0 | 0 | 67 | 6 | 36
days |  |  | 8 [5 to 18] | 6.5 [4.0 to 10.0] | 10 [4 to 22]

6. Secondary Outcome: Length of Hospitalization
Description: Duration of hospitalization
Time Frame: Day 1 through Day 30
Population: All subjects without mechanical ventilation- Part 2. Part 1 is designed as a randomized, double-blind, placebo-controlled, 3-arm, parallel-group study to evaluate the safety of plonmarlimab in subjects with severe COVID-19. So, no available efficacy data for this part.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- TJ003234 6mg/kg (Part 1): subjects treated with 6mg/kg
- TJ003234 6mg/kg (Part 2): subjects treated with 6 mg/kg TJ003234 (mITT population)
- TJ003234 10mg/kg (Part 2): subjects treated with 10mg/kg of TJ003234 (mITT population)
Arm/Group | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6mg/kg (Part 2) | TJ003234 10mg/kg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 0 | 0 | 67 | 6 | 36
days |  |  | 10 [8 to 13] | 9.5 [1 to 12] | 11 [7 to 18]

ADVERSE EVENTS:
Time Frame: All adverse events will be collected from the day of informed consent to Day 30.
Description: Disease progression or deterioration is also recorded as an AE/SAE, regardless of whether the Investigator assesses that it is related to the study drug. Signs and symptoms from the following may be considered AEs: drug overdose, withdrawal or misuse, drug interactions, extravasations, exposure during pregnancy/breastfeeding. Safety reporting results are based on ITT population.
Groups:
- TJ003234 3 mg/kg (Part 1): subjects treated with 3mg/kg TJ003234 (Part 1) (Safety population)
- TJ003234 6mg/kg (Part 1): subjects treated with 6 mg/kg TJ003234 (Safety population)
- Placebo (Part 1); Placebo (Part 2): subjects treated by placebo (Safety population)
- TJ003234 6 mg/kg (Part 2): subjects treated with 6mg/kg TJ003234 (Safety population)
- TJ003234 10mg/kg (Part 2): subjects treated with 10mg/kg (Safety population)
Arm/Group | TJ003234 3 mg/kg (Part 1) | TJ003234 6mg/kg (Part 1) | Placebo (Part 1) | TJ003234 6 mg/kg (Part 2) | TJ003234 10mg/kg (Part 2) | Placebo (Part 2)
All-Cause Mortality (participants affected / at risk) | 1/8 | 1/8 | 2/8 | 11/77 | 1/6 | 10/42
Serious Adverse Events (participants affected / at risk) | 2/8 | 4/8 | 2/8 | 22/77 | 1/6 | 16/42
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/77 | 0/6 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TJ003234 3 mg/kg (Part 1) (N=8) | TJ003234 6mg/kg (Part 1) (N=8) | Placebo (Part 1) (N=8) | TJ003234 6 mg/kg (Part 2) (N=77) | TJ003234 10mg/kg (Part 2) (N=6) | Placebo (Part 2) (N=42)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MYOCARDIAL ISCHEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WORSENING BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TAKOTSUBO CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MULTI ORGAN SYSTEM FAILURE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 4 (4)
BACTEREMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
(Worsening) PNEUMONIA (due to COVID-19) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
SELF-EXTUBATION WITH COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTRACRANIAL HEMORRHAGIC TRANSFORMATION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBARACHNOID HEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
(WORSENING) HYPOXIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (13) | 0 (0) | 5 (5)
(WORSENING) RESPIRATORY FAILURE DUE TO COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 4 (4)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WORSENING BILATERAL PNEUMONITITS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DISTRIBUTIVE SHOCK (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NECROTIC DIGITS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEMORRHAGIC SHOCK (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION WITH RAPID VENTRICULAR RESPONSE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MELENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HOSPITAL-ACQUIRED PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VENTILATOR ASSOCIATED PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 INDUCED MYOCARDITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AVULSION OF RIGHT COMMON FEMORAL ARTERY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE TUBULAR NECROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RIGHT AXILLARY DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERSISTENT SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endotracheal intubation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT04341116/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT04341116/SAP_001.pdf